CLINICAL TRIAL: NCT02947893
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Impact of Low Doses of Nilotinib (Tasigna®) on Safety, Biomarkers and Clinical Outcomes in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Impact of Nilotinib on Safety, Biomarkers and Clinical Outcomes in Mild to Moderate Alzheimer's Disease
Acronym: AD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, R. Scott Turner, Director, Memory Disorders Program, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-0315
Record Dates: First submitted 2016-10-21; First posted 2016-10-28 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer's Disease
Keywords: Nilotinib in Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — nilotinib; Amyloid beta-Protein Precursor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (placebo) (Placebo Comparator): Out of 42 total participants with mild to moderate AD (MMSE=17-24 inclusive) and their study partners that will be recruited and 1:1 randomized, 21 (twenty-one) will be assigned to group 1 and given 1 capsule of a placebo drug by mouth every day for the first 6 months followed by 2 capsules once daily for the subsequent 6 months, every time taken without a meal, for the total duration of the study for 12 months.
  Interventions: Drug: Placebo Capsule(s) Once a Day by Mouth
- Group 2 (treated) (Active Comparator): Out of 42 total participants with mild to moderate AD (MMSE=17-24 inclusive) and their study partners that will be recruited and 1:1 randomized, 21 (twenty-one) will be assigned to group 2 treated with 1 capsule (150mg Nilotinib) once a day by mouth for the first 6 months followed by dose escalation to 2 capsules (300mg Nilotinib) once daily by mouth for the subsequent 6 months, every time taken without a meal, for the total study duration of 12 months.
  Interventions: Drug: Nilotinib Capsule(s) Once a Day by Mouth

INTERVENTIONS:
Drug: Placebo Capsule(s) Once a Day by Mouth — 1 capsule of Placebo once a day for 6 months followed by 2 capsules of Placebo for another 6 months
  Other Names: Nilotinib in Alzheimer's Disease
  Arms: Group 1 (placebo)
Drug: Nilotinib Capsule(s) Once a Day by Mouth — 1 capsule of Nilotinib 150 mg once a day for 6 months followed by 2 capsules of Nilotinib (150 mg each capsule = 300 mb total) for the subsequent 6 months
  Other Names: Nilotinib in Alzheimer's Disease
  Arms: Group 2 (treated)

SUMMARY:
The investigators hypothesize that Nilotinib will be safe in individuals with mild to moderate AD. Specifically, investigators hypothesize that low daily oral doses of Nilotinib will lead to CSF penetration, CNS Abl inhibition, and stabilization of CSF total Tau and p-Tau231/181 and Abeta42/40 levels. The investigators hypothesize that Nilotinib will decrease brain load of amyloid using amyloid positron emission tomography (PET). The investigators also predict that Nilotinib will reduce CSF markers of cell death, including neuron specific enolase (NSE) and S100B.

DETAILED DESCRIPTION:
The investigators propose a novel treatment strategy that involves Abl inhibition to alter Abeta40/42, total Tau and p-Tau231/181 in subjects with mild to moderate dementia due to AD. The investigators pre-clinical studies show that Nilotinib inhibits brain Abl, decreases Abeta and p-Tau, modulates brain and peripheral immune profiles and reverses cognitive decline in AD models. Taken together, these data support the hypothesis that Nilotinib is a viable therapeutic candidate - via Abl inhibition - in subjects with AD. Based on strong pre-clinical evidence about the effects of Nilotinib on neurodegenerative pathologies, including autophagic clearance of neurotoxic proteins, immunity and behavior, the investigators conducted an open label pilot clinical trial in advanced (stage 3-5) PD with dementia (PDD) and Lewy Body Dementia (LBD) patients. Participants (N=12) were randomized 1:1 to once daily oral dose of 150mg and 300mg Nilotinib for 6 months. The investigators showed that Nilotinib penetrates the blood brain barrier (BBB), in agreement with pre-clinical data. Several studies show that Abeta42 is decreased and CSF total Tau and p-Tau are increased in PD and LBD. Investigators data show that Nilotinib reverses loss of CSF Abeta40/42 and significantly reduces (N=5, P<0.05) CSF total Tau and p-Tau between baseline and 6 months treatment. These biomarker changes are consistent with cognitive improvement (3.5-3.85 points) using Mini-Mental Status Exam (MMSE) and the Scales for Outcomes in Parkinson's Disease-Cognition (SCOPA-Cog) between baseline and 6 months. These data are very compelling to evaluate the effects of Nilotinib in a phase II, randomized, double-blind, placebo-controlled trial in patients with mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50
2. Fluent in English
3. Biomarker confirmed AD with CSF level of Abeta42 <600ng/mL
4. Able to ingest oral medications
5. Diagnosis of mild to moderate AD according to dementia criteria outlined by McKhann et al.
6. Neuroimaging (MRI or CT) consistent with the diagnosis of AD within the past year
7. MMSE between 17 and 24 (inclusive) at screening
8. Modified Hachinski score ≤ 4
9. QTc interval 350-460ms, inclusive
10. Caregiver/study partner to accompany participant to all visits and have direct contact with the participant > 2 days/week
11. Written informed consent
12. Capability and willingness to comply with all study criteria
13. Supervision available for study medication
14. Stable medical conditions for 3 months prior to screening visit
15. Stable medications for 4 weeks prior to screening visit
16. Able to complete baseline assessments
17. Minimum of 6 years of education, or work history sufficient to exclude mental retardation
18. Stable use of cholinesterase inhibitors and memantine (U.S. FDA-approved medications for patients with probable AD), vitamin E (up to 400 IU daily), estrogens, aspirin (81-300 mg daily), and cholesterol-lowering agents for 3 months prior to screening is allowed.
19. Clinical laboratory values within normal limits or, if abnormal, must be judged to be clinically insignificant by the investigator

Exclusion Criteria:

1. Non-AD dementia, probable AD with Down syndrome, APP, PS-1, or PS-2 mutations (known familial AD), LBD and Fronto-temporal dementia (FTD)
2. History of clinically significant stroke
3. Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
4. Sensory impairment that would preclude participation/cooperation with the protocol
5. Patients with hypokalemia, hypomagnesaemia, or long QTc syndrome.
6. Concomitant drugs known to prolong the QTc interval (>461ms) and history of cardiovascular disease, including myocardial infarction or cardiac failure, angina, arrhythmia
7. Prescribed strong CYP3A4 inhibitors or a medical history of liver or pancreatic disease
8. Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality
9. Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history of treated basal or squamous skin cancer, or stable prostate cancer are not exclusionary)
10. Pregnancy or possible pregnancy
11. Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder
12. Contraindication to MRI
13. Evidence of more than 4 micro hemorrhages and/or hemosiderosis by a recent (12 months) and/or the screening MRI.
14. A low B12 is exclusionary, unless follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant.
15. Enrolled in another active trial investigating an experimental drug or therapy for AD
16. HIV positive

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Safety will be measured by number of participants experiencing the occurrence of adverse events and/or abnormal laboratory values | 12 months
  Safety will be measured by assessing number of participants with abnormal laboratory values, as well as adverse events (AEs) and serious adverse events (SAEs) deemed to be possibly, probably, or definitely related to the study drug.

SECONDARY OUTCOMES:
Effects of Nilotinib treatment on measurement of Nilotinib in the CSF | 12 months
  The investigators will determine the effects of Nilotinib treatment on Abl inhibition to demonstrate CNS target engagement

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S. Turner, MD, PhD, Principal Investigator — Georgetown University; Charbel E Moussa, MD, PhD, Study Director — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pagan F, Hebron M, Valadez EH, Torres-Yaghi Y, Huang X, Mills RR, Wilmarth BM, Howard H, Dunn C, Carlson A, Lawler A, Rogers SL, Falconer RA, Ahn J, Li Z, Moussa C. Nilotinib Effects in Parkinson's disease and Dementia with Lewy bodies. J Parkinsons Dis. 2016 Jul 11;6(3):503-17. doi: 10.3233/JPD-160867. PMID 27434297
- See also: TRANSLATIONAL NEUROTHERAPEUTICS PROGRAM Georgetown University Medical Center & Medstar Georgetown University Hospital — https://neurology.georgetown.edu/translational_neurotherapeutics
- See also: Nilotinib - When the Hope outweighs the Hype — https://sites.google.com/a/georgetown.edu/moussa-lab/nilotinib---when-the-hope-outweighs-the-hype
- See also: The Laboratory for Dementia and Parkinsonism Georgetown University Medical Center — https://sites.google.com/a/georgetown.edu/moussa-lab/home